CLINICAL TRIAL: NCT02244281
Title: An Eight-week, Double-blind, Randomized, Parallel Group Design, Multicenter Study of FLOMAX® Capsules, 0.4 mg Daily Versus Placebo, in Female Patients With Lower Urinary Tract Symptoms (LUTS) With a Significant Component of Voiding Symptoms
Brief Title: Study of FLOMAX® Versus Placebo in Female Patients With Lower Urinary Tract Symptoms (LUTS) With a Significant Component of Voiding Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 527.25
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Lower Urinary Tract Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — Tamsulosin

ARMS (2):
- FLOMAX® (Experimental)
  Interventions: Drug: tamsulosin hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tamsulosin hydrochloride
  Other Names: FLOMAX®
  Arms: FLOMAX®
Drug: Placebo
  Arms: Placebo

SUMMARY:
1. To study the symptomatic improvement in LUTS afforded by FLOMAX® capsules, 0.4 mg daily compared to placebo, in female patients with lower urinary tract symptoms (LUTS) with a significant component of voiding symptoms
2. To study the improvement afforded by FLOMAX® capsules versus placebo, in this patient population, in quality of life
3. To assess the safety and tolerability of FLOMAX® capsules, 0.4 mg compared to placebo, in women suffering from LUTS with a significant component of voiding symptoms

ELIGIBILITY:
Inclusion Criteria:

* Adult women, 18 years of age or older, currently diagnosed with LUTS with a significant component of voiding symptoms
* The Patient must be diagnosed with one of the following: hesitancy, intermittency, difficulty in bladder emptying, or straining to void
* Patients must have had an AUA Symptom Score of 13 or higher
* Obstruction component of AUA Symptom Score (Items 1, 3, 5, and 6) had to be 5 points or higher
* Patients that are currently taking alpha-blockers or anticholinergics must discontinue the drugs at least 2 weeks prior to Visit 1
* Patients should show compliance of greater than or equal to 80% with placebo usage
* Patients should be surgically sterile, or 2 years postmenopausal, or practicing a medically acceptable method of birth control
* Patients must have a negative urine Beta Human Chorionic Gonadotropin (beta-HCG)
* Patients must be able to provide written informed consent prior to participation in the study in accordance with regulatory requirements
* Patients must be judged by the investigator to be reliable and should comply with all tests and examinations stipulated in the protocol
* All patients should be able to understand and read English

Exclusion Criteria:

* Patients who presented with an active urinary tract infection or who had presented with two or more culture positive urinary tract infections within 6 months of the study
* Patients with significant prolapse beyond the hymenal ring, per the investigator's judgment
* Patients who had taken anticholinergic medications for the treatment of other urologic conditions and had not discontinued their use 2 weeks prior to study entry
* Patients who had a history or active condition of renal or urethral calculi, urethral colic, mechanical outlet obstruction (i.e., bladder neck contracture or stricture, bladder tumor, or bladder calculi) 3 months prior to study entry
* Patients with a history of bladder, vaginal or urethral surgery in the last 6 months
* Patients who have a history of microscopic hematuria and not had a recent work-up including cystoscopy and upper urinary tract study (within 6 months of screening) or a diagnosis of a condition that may exclude the patient in the opinion of the investigator
* Abnormal urinalysis as defined by the following mid-stream, clean-catch specimen results:

  * A bacterial colony count of greater than 100,000/ml.
  * More than 10 leukocytes per high power field with more than two granular casts per high power field.
  * More than 10 red blood cells (non-menstrual tainted urine sample) per high power field.
  * Proteinuria >+1 (equivalent to >30 mg/dL)
* Patients presenting with any of the following: history of a neurogenic bladder due to any neurologic condition that might involve the lower urinary tract, active urinary stone disease, previous pelvic radiotherapy, perirectal inflammatory disorder or inflammatory bowel disease
* Patients that had a history of sexually transmitted diseases of the genitourinary system such as syphilis, herpes, gonorrhea, chlamydia, mycoplasma, trichomonas (within 3 months of the study) or any other diagnosis that in the opinion of the investigator may have excluded the patient
* Patients that are pregnant or breast-feeding
* The Patient has significant pelvic pain that demands treatment with narcotics
* Large fluctuations in LUTS symptoms over the last 6 months (i.e., symptoms appearing and disappearing with unusual rapidity)
* Any baseline (Visit 1) laboratory serum test with the following values: Hemoglobin: <11.0 g/dL, Leukocytes: <3,000 per mm3, Liver enzymes [serum glutamic oxaloacetic transaminase / Aspartate aminotransferase (SGOT/AST), serum glutamic pyruvic transaminase / Alanine transaminase (SGPT/ALT) or alkaline phosphatase]: more than two times the upper limit of normal at baseline (Visit 1). Serum creatinine more than two times the upper limit of normal at baseline (Visit 1)
* Patients with a diagnosis of cancer, except basal cell carcinoma, within the past 5 years. (Note: Contact the Trial Clinical Monitor with any specific or special circumstances regarding the entry of a cancer patient.)
* Participation in another drug study within 4 weeks of baseline (Visit 1)
* Clinically relevant conditions which may interfere with the patient's ability to participate in the study including, but not limited to, the following: neurologic, gastrointestinal, cardiovascular, hepatic, renal, psychiatric, hematologic or respiratory disease and clinically relevant laboratory abnormalities not mentioned above (e.g., hematuria) based upon the clinical judgment of the investigator
* Patients who have been receiving cimetidine, ranitidine and warfarin medications within 2 weeks of screening and who would potentially use such medication during the course of the trial
* Patients with known hypersensitivity to FLOMAX® (tamsulosin hydrochloride) or other alpha-blockers
* Patients with a history of myocardial infarction within 6 months of baseline (Visit 1)
* Patients with uncontrolled hypertension (systolic >160 mmHg, diastolic >100 mmHg) and patients with severe hypotension (systolic <90 mmHg) after 5 minutes of sitting
* Patients who have been using the following drugs, within 2 weeks prior to screening (Visit 1), and who are unable to discontinue these drugs over the course of the study

  1. Alpha-adrenergic blocking agents
  2. Alpha-adrenergic medication
  3. Drugs with systemic anticholinergic activity including antihistamines. Antihistamines allowed are Allegra®, Claritin® and Zyrtec®
  4. Antispasmodics or muscle relaxants
  5. Parasympathomimetics, cholinomimetics, and/or similar drugs
* Patients with poorly controlled diabetes mellitus based upon urine with 2+ (or greater) glucose on urinalysis, performed at screening (Visit 1).
* Patients who suffer from neurological diseases affecting the bladder (i.e., multiple sclerosis, Parkinson's disease, stroke, and any bladder trauma that may have been an exclusion criterion in the opinion of the investigator)
* Patients that have a neurological impairment or psychiatric disorder that prevents their comprehension of consent and their ability to comply with the protocol
* Patients who had been diagnosed with interstitial cystitis according to the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) criteria
* Patients that had a history of urethral syndrome whose treatment was other than dilation. Patients treated by dilation 3 months prior to study entry were allowed to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2001-05; Primary Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Assessment of efficacy on a American Urological Association (AUA) Symptom Score Index | Up to day 56 after first study drug administration

SECONDARY OUTCOMES:
Assessment of Quality of Life on a incontinence impact questionary and urogenital distress inventory | Up to day 56 after first study drug administration
Assessment of urinary frequency and nocturia on a seventy-two hour voiding diary | Up to day 28 after first study drug administration
Assessment of urinary obstruction | Up to day 56 after first study drug administration
  by uroflowmetry
Assessment of Post-Void Residual volume | Up to day 56 after first study drug administration
  by pelvic ultrasound
Assessment of lower urinary tract symptoms of obstruction | Up to day 56 after first study drug administration
  (voiding, Items 1, 3, 5 and 6), irritation (storage, Items 2, 4 and 7) and nocturia (Item 7) by AUA Symptom Score Index sub scores
Number of patients with adverse events | Up to day 56 after first study drug administration